CLINICAL TRIAL: NCT02357303
Title: Premedication With Simethicone and N-acetylcysteine in Improving Mucosal Visibility During Upper Endoscopy - a Prospective Double-blinded Randomized Controlled Trial
Brief Title: Simethicone and N-acetylcysteine in Upper Endoscopy - Prospective Double-blinded Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Portuguese Oncology Institute, Coimbra (Other)
Responsible Party: Principal Investigator, Luís André Caio Elvas, Principal Investigator, Portuguese Oncology Institute, Coimbra
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: PortugueseOIC 001
Record Dates: First submitted 2015-01-29; First posted 2015-02-06 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Gastric Mucosal Lesion
Keywords: Randomized controlled trial; Endoscopy; Gastric mucosa; Simethicone; Acetylcysteine
MeSH Terms: interventions — Simethicone; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Group A - 100mL of water by mouth, 15 to 30 minutes before endoscopy
  Interventions: Other: Placebo
- Simethicone (Active Comparator): Group B - 100mL of water plus 100mg Simethicone by mouth, 15 to 30 minutes before endoscopy
  Interventions: Drug: Simethicone
- Simethicone plus N-acetylcysteine (Active Comparator): Group C - 100mL of water plus 100mg Simethicone plus 600mg N-acetylcysteine by mouth, 15 to 30 minutes before endoscopy
  Interventions: Drug: Acetylcysteine

INTERVENTIONS:
Drug: Simethicone — 100mL of water plus 100mg Simethicone by mouth, 15 to 30 minutes before endoscopy
  Other Names: Aero-OM
  Arms: Simethicone
Drug: Acetylcysteine — 100mL of water plus 100mg Simethicone plus 600mg N-acetylcysteine by mouth, 15 to 30 minutes before endoscopy
  Other Names: Fluimucil
  Arms: Simethicone plus N-acetylcysteine
Other: Placebo — 100mL of water
  Arms: Placebo

SUMMARY:
The upper endoscopy is one of the most common methods for the diagnosis and treatment of upper gastrointestinal (GI) tract diseases and provides a unique opportunity to identify early neoplastic lesions.

Before an upper endoscopy it is required a 6 hour fasting period[1]. However, even with this fasting period, sometimes the mucosal visualization, especially in the stomach, is impaired by the presence of foam, bubbles or gastric mucus.

To improve visualization of the gastric mucosa, it is possible to administrate an oral solution of defoaming agents such as Simethicone and mucolytic agents like Pronase or N-Acetylcysteine previously to the procedure.

The aim of this project is to determine if the use of premedication with simethicone, alone or in association with N-Acetylcysteine, improves mucosal visualization during an upper GI endoscopy.

DETAILED DESCRIPTION:
a. Study type: prospective, randomized, double-blinded, placebo-controlled trial: i. Prospective inclusion of patients; ii. Randomization by computer generated tables; iii. Allocation concealment by sealed, opaque envelopes; iv. Double-blinded - nurse instructed not to reveal treatment; patient and doctor unaware of treatment;

b. Patient selection: consecutive series of patients scheduled for upper gastrointestinal endoscopy; Exclusion criteria - sedation, previous total gastrectomy, known neoplasia or stenosis, allergies to simethicone or N-acetylcysteine, therapeutic or urgent procedures;

c. Sample size: 270 (3 groups of 90 patients): to improve "excellent" preparations from 20% (value from our own database) to 40% and assuming a normal distribution and a power of 80% (α=0.05), the calculated sample size of each of the 3 groups was 82; allowing for a 10% dropout rate, the sample size is 90 (270 patients overall); Groups: Group A - 100mL of water (placebo); Group B - 100mL of water plus 100mg Simethicone; Group C - 100mL of water plus 100mg Simethicone plus 600mg N-acetylcysteine;

d. Data collection methods: form sheet filled by nurses (appendix 1) and endoscopist (appendix 2);

e. Analysed variables: patients characteristics (age, gender), indication for endoscopy, time from administration to procedure, score of mucosal visualization, side effects of medication;

f. Statistical analysis: chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* consecutive series of patients scheduled for upper gastrointestinal endoscopy
* signed informed consent

Exclusion Criteria:

* sedation
* previous total gastrectomy
* known neoplasia or stenosis
* therapeutic or urgent procedures
* allergies to simethicone or N-acetylcysteine

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Score of mucosal visualization | 1 day (During endoscopy)
  Evaluation of the visibility of gastric mucosa during upper endoscopy using a scale (excelent, adequadate or inadequate) for esophagus, stomach and duodenum

OTHER OUTCOMES:
Drug side effects | 1 day (During endoscopy)
  Evaluation of the drug side effects during upper endoscopy (report of any allergic reaction)

CONTACTS AND LOCATIONS:
Overall Officials: Luís Elvas, MD, Principal Investigator — Gastroenterology Department, Portuguese Oncology Institute - Coimbra
Locations (1):
- Portuguese Oncology Institute - Coimbra, Coimbra, Coimbra District, Portugal

REFERENCES:
- [Background] Faigel DO, Eisen GM, Baron TH, Dominitz JA, Goldstein JL, Hirota WK, Jacobson BC, Johanson JF, Leighton JA, Mallery JS, Raddawi HM, Vargo JJ 2nd, Waring JP, Fanelli RD, Wheeler-Harbough J; Standards of Practice Committee. American Society for Gastrointestinal Endoscopy. Preparation of patients for GI endoscopy. Gastrointest Endosc. 2003 Apr;57(4):446-50. doi: 10.1016/s0016-5107(03)80006-8. No abstract available. PMID 12665751
- [Background] Asl SM, Sivandzadeh GR. Efficacy of premedication with activated Dimethicone or N-acetylcysteine in improving visibility during upper endoscopy. World J Gastroenterol. 2011 Oct 7;17(37):4213-7. doi: 10.3748/wjg.v17.i37.4213. PMID 22072853
- [Background] Chen MJ, Wang HY, Chang CW, Hu KC, Hung CY, Chen CJ, Shih SC. The add-on N-acetylcysteine is more effective than dimethicone alone to eliminate mucus during narrow-band imaging endoscopy: a double-blind, randomized controlled trial. Scand J Gastroenterol. 2013 Feb;48(2):241-5. doi: 10.3109/00365521.2012.749509. Epub 2012 Dec 27. PMID 23268593
- [Background] Bhandari P, Green S, Hamanaka H, Nakajima T, Matsuda T, Saito Y, Oda I, Gotoda T. Use of Gascon and Pronase either as a pre-endoscopic drink or as targeted endoscopic flushes to improve visibility during gastroscopy: a prospective, randomized, controlled, blinded trial. Scand J Gastroenterol. 2010 Mar;45(3):357-61. doi: 10.3109/00365520903483643. PMID 20148732
- [Background] Ahsan M, Babaei L, Gholamrezaei A, Emami MH. Simethicone for the Preparation before Esophagogastroduodenoscopy. Diagn Ther Endosc. 2011;2011:484532. doi: 10.1155/2011/484532. Epub 2011 Aug 4. PMID 21826120
- [Background] Bertoni G, Gumina C, Conigliaro R, Ricci E, Staffetti J, Mortilla MG, Pacchione D. Randomized placebo-controlled trial of oral liquid simethicone prior to upper gastrointestinal endoscopy. Endoscopy. 1992 May;24(4):268-70. doi: 10.1055/s-2007-1010479. PMID 1612040
- [Background] Keeratichananont S, Sobhonslidsuk A, Kitiyakara T, Achalanan N, Soonthornpun S. The role of liquid simethicone in enhancing endoscopic visibility prior to esophagogastroduodenoscopy (EGD): A prospective, randomized, double-blinded, placebo-controlled trial. J Med Assoc Thai. 2010 Aug;93(8):892-7. PMID 20718163
- [Background] Kuo CH, Sheu BS, Kao AW, Wu CH, Chuang CH. A defoaming agent should be used with pronase premedication to improve visibility in upper gastrointestinal endoscopy. Endoscopy. 2002 Jul;34(7):531-4. doi: 10.1055/s-2002-33220. PMID 12170403
- [Background] Lee GJ, Park SJ, Kim SJ, Kim HH, Park MI, Moon W. Effectiveness of Premedication with Pronase for Visualization of the Mucosa during Endoscopy: A Randomized, Controlled Trial. Clin Endosc. 2012 Jun;45(2):161-4. doi: 10.5946/ce.2012.45.2.161. Epub 2012 Jun 30. PMID 22866258
- [Background] Fujii T, Iishi H, Tatsuta M, Hirasawa R, Uedo N, Hifumi K, Omori M. Effectiveness of premedication with pronase for improving visibility during gastroendoscopy: a randomized controlled trial. Gastrointest Endosc. 1998 May;47(5):382-7. doi: 10.1016/s0016-5107(98)70223-8. PMID 9609431
- [Background] Zala G, Flury R, Wust J, Meyenberger C, Ammann R, Wirth HP. [Omeprazole/amoxicillin: improved eradication of Helicobacter pylori in smokers because of N-acetylcysteine]. Schweiz Med Wochenschr. 1994 Aug 9;124(31-32):1391-7. German. PMID 8091167
- [Background] Chang CC, Chen SH, Lin CP, Hsieh CR, Lou HY, Suk FM, Pan S, Wu MS, Chen JN, Chen YF. Premedication with pronase or N-acetylcysteine improves visibility during gastroendoscopy: an endoscopist-blinded, prospective, randomized study. World J Gastroenterol. 2007 Jan 21;13(3):444-7. doi: 10.3748/wjg.v13.i3.444. PMID 17230616
- [Background] Chang WK, Yeh MK, Hsu HC, Chen HW, Hu MK. Efficacy of simethicone and N-acetylcysteine as premedication in improving visibility during upper endoscopy. J Gastroenterol Hepatol. 2014 Apr;29(4):769-74. doi: 10.1111/jgh.12487. PMID 24325147
- [Derived] Elvas L, Areia M, Brito D, Alves S, Saraiva S, Cadime AT. Premedication with simethicone and N-acetylcysteine in improving visibility during upper endoscopy: a double-blind randomized trial. Endoscopy. 2017 Feb;49(2):139-145. doi: 10.1055/s-0042-119034. Epub 2016 Nov 16. PMID 27852098